CLINICAL TRIAL: NCT00348998
Title: Pilot Phase II Trial of Bevacizumab in Combination With Hormonal and Radiotherapy in Patients With High-Risk Prostate Cancer
Brief Title: Bevacizumab, Hormone Therapy, and Radiation Therapy in Treating Patients With Locally Advanced Prostate Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Virginia Mason Hospital/Medical Center (Other)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000480370; BRIVMRC-3031500; GENENTECH-AVF3549s
Record Dates: First submitted 2006-07-05; First posted 2006-07-06 (Estimated); Last update posted 2013-11-06 (Estimated); Status verified 2008-11

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; stage IIB prostate cancer; stage IIA prostate cancer; stage III prostate cancer; stage IV prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Bevacizumab; bicalutamide; Goserelin; Radiotherapy

INTERVENTIONS:
Biological: bevacizumab
Drug: bicalutamide
Drug: goserelin acetate
Radiation: radiation therapy

SUMMARY:
RATIONALE: Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Androgens can cause the growth of prostate cancer cells. Drugs, such as goserelin and bicalutamide, may stop the adrenal glands from making androgens. Radiation therapy uses high-energy x-rays to kill tumor cells. Bevacizumab may also make tumor cells more sensitive to radiation therapy. Giving bevacizumab together with hormone therapy and radiation therapy may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving bevacizumab together with hormone therapy and radiation therapy works in treating patients with high-risk locally advanced prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the safety and efficacy of giving bevacizumab together with hormonal therapy and radiotherapy in patients with high-risk locally advanced prostate cancer.

OUTLINE: This is an open-label, pilot study.

Beginning in week 1, patients receive goserelin subcutaneously once every 3 months for 2 years. Patients also receive oral bicalutamide once daily and bevacizumab IV over 30- to 90-minutes once every 2 weeks in weeks 1-16 and undergo radiotherapy 5 days a week in weeks 9-16. After completion of radiotherapy, patients receive a higher dose of bevacizumab once every 3 weeks in weeks 17-28.

After completion of study treatment, patients are evaluated at 30 days.

PROJECTED ACCRUAL: A total of 18 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the prostate

  * High-risk, locally advanced disease (T2b-T4 disease), meeting 1 of the following criteria:

    * Gleason score 8-10
    * Prostate-specific antigen > 20 ng/dL AND Gleason score 7

      * T2a disease allowed provided ≥ 5 biopsies contain Gleason score 4 +3 cancer (minimum of 10 biopsies total required)
* No evidence of metastatic disease within the past 60 days by physical examination, chest x-ray, bone scan, and CT scan of abdomen and pelvis

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Hemoglobin > 8 g/dL
* Absolute granulocyte count ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* Creatinine ≤ 1.5 times ULN
* Blood pressure ≤ 150/100 mm Hg
* No cardiovascular disease, including any of the following:

  * Unstable angina
  * New York Heart Association class II-IV congestive heart failure
  * History of myocardial infarction within the past 6 months
  * History of stroke within the past 6 months

PRIOR CONCURRENT THERAPY:

* At least 4 weeks since prior major surgery
* No prior hormonal therapy (except finasteride for obstructive voiding symptoms) for prostate cancer
* No prior or concurrent chemotherapy, biologic therapy, or radiotherapy for prostate cancer

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2006-04

PRIMARY OUTCOMES:
Safety
Efficacy

CONTACTS AND LOCATIONS:
Overall Officials: Jacqueline Vuky, MD, Study Chair — Virginia Mason Hospital/Medical Center
Locations (1):
- Benaroya Research Institute at Virginia Mason Medical Center, Seattle, Washington, United States

REFERENCES:
- [Background] Karlou M, Tzelepi V, Efstathiou E. Therapeutic targeting of the prostate cancer microenvironment. Nat Rev Urol. 2010 Sep;7(9):494-509. doi: 10.1038/nrurol.2010.134. PMID 20818327